CLINICAL TRIAL: NCT00996580
Title: A Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of a Combination Oral Contraceptive Regimen (DR-103) for the Prevention of Pregnancy in Women
Brief Title: A Study to Evaluate the Efficacy and Safety of DR-103 for the Prevention of Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Women's Health (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DR-103-301
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2013-06-14 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Pregnancy Prevention
Keywords: Contraception; Oral contraceptives
MeSH Terms: interventions — HLA-DR103 antigen; Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DR-103 (Experimental): Four 91-day cycles of the DR-103 regimen:
  * 42 days combination therapy of 20 mcg ethinyl estradiol (EE) /150 mcg levonorgestrel (LNG) followed by;
  * 21 days combination therapy of 25 mcg EE/150 mcg LNG followed by;
  * 21 days combination therapy of 30 mcg EE/150 mcg LNG followed by;
  * 7 days of 10 mcg EE.
  Interventions: Drug: DR-103

INTERVENTIONS:
Drug: DR-103 — One tablet daily.
  Four 91-day cycles of the DR-103 regimen:
  42 days combination therapy of 20 mcg ethinyl estradiol (EE) /150 mcg levonorgestrel (LNG) followed by; 21 days combination therapy of 25 mcg EE/150 mcg LNG followed by; 21 days combination therapy of 30 mcg EE/150 mcg LNG followed by; 7 days of 10 mcg EE.
  Other Names: levonorgestrel/ethinyl estradiol; Quartette®

SUMMARY:
This is an open-label, single-treatment study. All subjects will receive 12 months of oral contraceptive therapy with DR-103. Study participants will receive physical and gynecological exams, including Pap smear. During the study, all participants will be required to complete a diary.

ELIGIBILITY:
Inclusion Criteria:

* Sexually active at risk for pregnancy
* Agreement to use study OC therapy as their only method of birth control during the study
* history of regular spontaneous menstrual cycles or withdrawal bleeding episodes
* Others as dictated by FDA-approved protocol

Exclusion Criteria:

* Any contraindication to the use of oral contraceptives
* Pregnancy or plans to become pregnant in the next 14 months
* Smoker and age ≥ 35 years
* Others as dictated by FDA-approved protocol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3597 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (86):
- United States (86):
  - Teva Women's Health Research Investigational Site, Montgomery, Alabama
  - Teva Women's Health Research Investigational Site, Phoenix, Arizona
  - Teva Women's Health Research Investigational Site, Tucson, Arizona
  - Teva Women's Health Research Investigational Site, Little Rock, Arkansas
  - Teva Women's Health Research Investigational Site, Anaheim, California
  - Teva Women's Health Research Investigational Site, Irvine, California
  - Teva Women's Health Research Investigational Site, Los Angeles, California
  - Teva Women's Health Research Investigational Site, National City, California
  - Teva Women's Health Research Investigational Site, San Diego, California
  - Teva Women's Health Research Investigational Site, San Francisco, California
  - Teva Women's Health Research Investigational Site, Torrance, California
  - Teva Women's Health Research Investigational Site, Colorado Springs, Colorado
  - Teva Women's Health Research Investigational Site, Pueblo, Colorado
  - Teva Women's Health Research Investigational Site, Washington D.C., District of Columbia
  - Teva Women's Health Research Investigational Site, Clearwater, Florida
  - Teva Women's Health Research Investigational Site, Jacksonville, Florida
  - Teva Women's Health Research Investigational Site, Leesburg, Florida
  - Teva Women's Health Research Investigational Site, Miami, Florida
  - Teva Women's Health Research Investigational Site, New Port Richey, Florida
  - Teva Women's Health Research Investigational Site, Palm Beach, Florida
  - Teva Women's Health Research Investigational Site, St. Petersburg, Florida
  - Teva Women's Health Research Investigational Site, Tampa, Florida
  - Teva Women's Health Research Investigational Site, West Palm Beach, Florida
  - Teva Women's Health Research Investigational Site, Atlanta, Georgia
  - Teva Women's Health Research Investigational Site, Decatur, Georgia
  - Teva Women's Health Research Investigational Site, Roswell, Georgia
  - Teva Women's Health Research Investigational Site, Sandy Springs, Georgia
  - Teva Women's Health Research Investigational Site, Savannah, Georgia
  - Teva Women's Health Research Investigational Site, Meridian, Idaho
  - Teva Women's Health Research Investigational Site, Champaign, Illinois
  - Teva Women's Health Research Investigational Site, Wichita, Kansas
  - Teva Women's Health Research Investigational Site, Lexington, Kentucky
  - Teva Women's Health Research Investigational Site, Louisville, Kentucky
  - Teva Women's Health Research Investigational Site, Mount Sterling, Kentucky
  - Teva Women's Health Research Investigational Site, Baton Rouge, Louisiana
  - Teva Women's Health Research Investigational Site, Metairie, Louisiana
  - Teva Women's Health Research Investigational Site, Baltimore, Maryland
  - Teva Women's Health Research Investigational Site, Kansas City, Missouri
  - Teva Women's Health Research Investigational Site, St Louis, Missouri
  - Teva Women's Health Research Investigational Site, Lincoln, Nebraska
  - Teva Women's Health Research Investigational Site, Las Vegas, Nevada
  - Teva Women's Health Research Investigational Site, Berlin, New Jersey
  - Teva Women's Health Research Investigational Site, Lawrenceville, New Jersey
  - Teva Women's Health Research Investigational Site, Moorestown, New Jersey
  - Teva Women's Health Research Investigational Site, New Brunswick, New Jersey
  - Teva Women's Health Research Investigational Site, Albuquerque, New Mexico
  - Teva Women's Health Research Investigational Site, Port Jefferson, New York
  - Teva Women's Health Research Investigational Site, Rochester, New York
  - Teva Women's Health Research Investigational Site, Cary, North Carolina
  - Teva Women's Health Research Investigational Site, Charlotte, North Carolina
  - Teva Women's Health Research Investigational Site, New Bern, North Carolina
  - Teva Women's Health Research Investigational Site, Raleigh, North Carolina
  - Teva Women's Health Research Investigational Site, Salisbury, North Carolina
  - Teva Women's Health Research Investigational Site, Wilmington, North Carolina
  - Teva Women's Health Research Investigational Site, Winston-Salem, North Carolina
  - Teva Women's Health Research Investigational Site, Columbus, Ohio
  - Teva Women's Health Research Investigational Site, Edmond, Oklahoma
  - Teva Women's Health Research Investigational Site, Oklahoma City, Oklahoma
  - Teva Women's Health Research Investigational Site, Eugene, Oregon
  - Teva Women's Health Research Investigational Site, Medford, Oregon
  - Teva Women's Health Research Investigational Site, Philadelphia, Pennsylvania
  - Teva Women's Health Research Investigational Site, Pittsburgh, Pennsylvania
  - Teva Women's Health Research Investigational Site, Charleston, South Carolina
  - Teva Women's Health Research Investigational Site, Columbia, South Carolina
  - Teva Women's Health Research Investigational Site, Goose Creek, South Carolina
  - Teva Women's Health Research Investigational Site, Greenville, South Carolina
  - Teva Women's Health Research Investigational Site, Greer, South Carolina
  - Teva Women's Health Research Investigational Site, Hilton Head Island, South Carolina
  - Teva Women's Health Research Investigational Site, Bristol, Tennessee
  - Teva Women's Health Research Investigational Site, Jackson, Tennessee
  - Teva Women's Health Research Investigational Site, Knoxville, Tennessee
  - Teva Women's Health Research Investigational Site, Memphis, Tennessee
  - Teva Women's Health Research Investigational Site, Nashville, Tennessee
  - Teva Women's Health Research Investigational Site, Austin, Texas
  - Teva Women's Health Research Investigational Site, Dallas, Texas
  - Teva Women's Health Research Investigational Site, Fort Worth, Texas
  - Teva Women's Health Research Investigational Site, Houston, Texas
  - Teva Women's Health Research Investigational Site, San Antonio, Texas
  - Teva Women's Health Research Investigational Site, Waco, Texas
  - Teva Women's Health Research Investigational Site, Salt Lake City, Utah
  - Teva Women's Health Research Investigational Site, Arlington, Virginia
  - Teva Women's Health Research Investigational Site, Newport News, Virginia
  - Teva Women's Health Research Investigational Site, Norfolk, Virginia
  - Teva Women's Health Research Investigational Site, Richmond, Virginia
  - Teva Women's Health Research Investigational Site, Seattle, Washington
  - Teva Women's Health Research Investigational Site, Tacoma, Washington

REFERENCES:
- [Result] Poindexter A, Reape KZ, Hait H. Efficacy and safety of a 28-day oral contraceptive with 7 days of low-dose estrogen in place of placebo. Contraception. 2008 Aug;78(2):113-9. doi: 10.1016/j.contraception.2008.04.001. Epub 2008 Jun 2. PMID 18672111
- [Derived] Portman DJ, Kaunitz AM, Howard B, Weiss H, Hsieh J, Ricciotti N. Efficacy and safety of an ascending-dose, extended-regimen levonorgestrel/ethinyl estradiol combined oral contraceptive. Contraception. 2014 Apr;89(4):299-306. doi: 10.1016/j.contraception.2014.01.013. Epub 2014 Jan 29. PMID 24576794

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 4,962 subjects were screened for participation in this study, and 3,597 took at least one dose of investigational product (Safety population).
Period: Overall Study
Arm/Group | DR-103
Started | 3597
Pregnancy Intent-to-Treat Population | 3019
Completed | 2144
Not Completed | 1453
Not completed — Adverse Event | 466
Not completed — Lost to Follow-up | 480
Not completed — Noncompliance with the protocol | 137
Not completed — Physician Decision | 5
Not completed — Pregnancy | 68
Not completed — Protocol Violation | 16
Not completed — Sponsor requested participant withdrawal | 35
Not completed — Withdrawal by Subject | 217
Not completed — Other | 29

BASELINE CHARACTERISTICS:
Population: Safety population: participants who took at least one dose of intervention.
Arm/Group | DR-103
Number analyzed (Participants) | 3597
Age Continuous [Mean (Standard Deviation); unit: years] | 27.4 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3597
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 14
  Asian | 78
  Native Hawaiian or Other Pacific Islander | 10
  Black or African American | 696
  White | 2324
  Hispanic or Latino | 404
  Other | 71
Height [Mean (Standard Deviation); unit: inches] | 64.6 (2.7)
Weight [Mean (Standard Deviation); unit: pounds] | 162.5 (43.2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (7.0)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 113.1 (10.4)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 72.3 (8.3)
Heart Rate [Mean (Standard Deviation); unit: beats/minute] | 74.6 (10.0)
Oral Contraceptive Use History [Number; unit: participants]
  Continuous user | 1570
  New Start | 619
  Prior User | 1408
Smoking Status [Number; unit: participants]
  Current Smoker | 602
  Former Smoker | 636
  Never Smoked | 2359

OUTCOME MEASURES:

1. Primary Outcome: All Users Pregnancy Rates Based on Pearl Index (PI) Analyses for 91-Day Cycles and Broken Out by Subpopulations Defined by Participant Weight
Description: Contraceptive failure is measured by the pregnancy rate calculated using the Pearl Index (PI). PI used all pregnancies, as determined by a positive urine and/or serum pregnancy test, except those for which the date of conception was before starting DR-103 or > 7 days after stopping the combination EE/LNG treatment of DR-103. The estimated date of conception and gestational age of the fetus was determined by transvaginal or abdominal ultrasound.
  The PI is defined as number of contraceptive failures per 100 women-years of exposure:
  (100)*(total number of pregnancies)*(4)/(total number of 91-day cycles)
Time Frame: Day 1 up to year 1
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age when study treatment started. The 'All Users' set included PITT participants who completed at least one 91-day cycle.
Measure: Number (95% Confidence Interval); unit: pregnancies / 100 woman years exposure
Units Other Than Participants: Treatment cycles
Groups:
- DR-103: Total: Four 91-day cycles of the DR-103 regimen:
  * 42 days combination therapy of 20 mcg ethinyl estradiol (EE) /150 mcg levonorgestrel (LNG) followed by;
  * 21 days combination therapy of 25 mcg EE/150 mcg LNG followed by;
  * 21 days combination therapy of 30 mcg EE/150 mcg LNG followed by;
  * 7 days of 10 mcg EE.
- DR-103: <90 kg Subpopulation: Subpopulation of the total participants who weighed <90 kg during the screening visit.
- DR-103: >=90kg Subpopulation: Subpopulation of the total participants who weighed >=90 kg during the screening visit.
Arm/Group | DR-103: Total | DR-103: <90 kg Subpopulation | DR-103: >=90kg Subpopulation
Number analyzed (Participants) | 2769 | 2276 | 493
Number analyzed (Treatment cycles) | 9217 | 7633 | 1584
pregnancies / 100 woman years exposure | 2.82 [2.1787 to 3.5920] | 2.46 [1.8111 to 3.2719] | 4.54 [2.6963 to 7.1601]

2. Primary Outcome: Typical-Use Pregnancy Rates Based on Pearl Index (PI) Analyses for 91-Day Cycles and Broken Out by Subpopulations Defined by Participant Weight
Description: as for outcome 1
Time Frame: Day 1 up to year 1
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age when study treatment started. The 'Typical-Use' set included PITT participants who completed at least one 91-day cycle and no other birth control methods including condoms were used.
Measure: Number (95% Confidence Interval); unit: pregnancies / 100 woman years exposure
Arm/Group | DR-103: Total | DR-103: <90 kg Subpopulation | DR-103: >=90kg Subpopulation
Number analyzed (Participants) | 2606 | 2149 | 457
pregnancies / 100 woman years exposure | 3.25 [2.5101 to 4.1372] | 2.83 [2.0793 to 3.7556] | 5.32 [3.1636 to 8.3840]

3. Primary Outcome: Compliant-Use Pregnancy Rates Based on Pearl Index (PI) Analyses for 91-Day Cycles and Broken Out by Subpopulations Defined by Participant Weight
Description: as for outcome 1
Time Frame: Day 1 up to year 1
Population: 'Compliant-Use' set included PITT participants who completed at least one 91-day cycle and no other birth control methods were used. Cycles were excluded if a subject 1) skipped 2 or more consecutive combination pills, 2) had a pattern of substantial non-compliance with treatment, or 3) used a prohibited concomitant medication
Measure: Number (95% Confidence Interval); unit: pregnancies / 100 woman years exposure
Arm/Group | DR-103: Total | DR-103: <90 kg Subpopulation | DR-103: >=90kg Subpopulation
Number analyzed (Participants) | 2505 | 2067 | 438
pregnancies / 100 woman years exposure | 3.71 [2.8629 to 4.7173] | 3.23 [2.3742 to 4.2869] | 6.04 [3.5894 to 9.5044]

4. Secondary Outcome: All Users Life-Table Estimates of Pregnancy Rates Based on 91-day Cycles and Broken Out by Subpopulations Defined by Participant Weight
Description: A life table approach was used to estimate the cumulative pregnancy rate on a cycle-by-cycle basis for each of the four 91-day treatment cycles.
Time Frame: Day 1 up to year 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: pregnancies / cumulative exposure
Arm/Group | DR-103: Total | DR-103: <90 kg Subpopulation | DR-103: >=90kg Subpopulation
Number analyzed (Participants) | 2769 | 2276 | 493
pregnancies / cumulative exposure
  Cycle 1 | 0.0074 [0.0048 to 0.0113] | 0.0060 [0.0035 to 0.0101] | 0.0139 [0.0066 to 0.0289]
  Cycle 2 | 0.0134 [0.0097 to 0.0186] | 0.0114 [0.0077 to 0.0168] | 0.0231 [0.0129 to 0.0415]
  Cycle 3 | 0.0212 [0.0162 to 0.0277] | 0.0185 [0.0135 to 0.0254] | 0.0339 [0.0205 to 0.0558]
  Cycle 4 | 0.0272 [0.0213 to 0.0346] | 0.0239 [0.0179 to 0.0317] | 0.0429 [0.0270 to 0.0676]

5. Primary Outcome: All Users Pregnancy Rates Based on Pearl Index (PI) Analyses for 28-Day Cycle-Equivalents and Broken Out by Subpopulations Defined by Participant Weight
Description: Contraceptive failure is measured by the pregnancy rate calculated using the Pearl Index (PI). PI used all pregnancies, as determined by a positive urine and/or serum pregnancy test, except those for which the date of conception was before starting DR-103 or > 7 days after stopping the combination EE/LNG treatment of DR-103. The estimated date of conception and gestational age of the fetus was determined by transvaginal or abdominal ultrasound.
  In order to compare the efficacy of extended treatment with DR-103 to conventional 28-day cyclic oral contraceptive treatment, the 91-day DR-103 treatment cycle was separated into three 28-day cycle-equivalents, derived from the 84-day active combination (EE/LNG) pill period of each 91-day extended cycle.
  The PI is defined as number of contraceptive failures per 100 women-years of exposure:
  (100)*(total number of pregnancies)*(13)/(total number of 28-day cycles)
Time Frame: Day 1 up to year 1
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age when study treatment started. The 'All Users' set included PITT participants who completed at least one 28-day cycle.
Measure: Number (95% Confidence Interval); unit: pregnancies / 100 woman years exposure
Units Other Than Participants: Treatment cycles
Arm/Group | DR-103: Total | DR-103: <90 kg Subpopulation | DR-103: >=90kg Subpopulation
Number analyzed (Participants) | 3019 | 2479 | 540
Number analyzed (Treatment cycles) | 30785 | 25487 | 5298
pregnancies / 100 woman years exposure | 2.74 [2.1189 to 3.4975] | 2.40 [1.7618 to 3.1869] | 4.42 [2.6192 to 6.9735]

6. Primary Outcome: Typical-Use Pregnancy Rates Based on Pearl Index (PI) Analyses for 28-Day Cycle-Equivalents and Broken Out by Subpopulations Defined by Participant Weight
Description: as for outcome 5
Time Frame: Day 1 up to year 1
Population: Pregnancy Intent-to-Treat Population (PITT) of participants who were 18 to 35 years of age when study treatment started. The 'Typical-Use' set included PITT participants who completed at least one 28-day cycle and no other birth control methods including condoms were used.
Measure: Number (95% Confidence Interval); unit: pregnancies / 100 woman years exposure
Arm/Group | DR-103: Total | DR-103: <90 kg Subpopulation | DR-103: >=90kg Subpopulation
Number analyzed (Participants) | 2972 | 2436 | 536
pregnancies / 100 woman years exposure | 2.92 [2.2558 to 3.7234] | 2.55 [1.8745 to 3.3905] | 4.72 [2.7973 to 7.4467]

7. Primary Outcome: Compliant-Use Pregnancy Rates Based on Pearl Index (PI) Analyses for 28-Day Cycle-Equivalents and Broken Out by Subpopulations Defined by Participant Weight
Description: as for outcome 5
Time Frame: Day 1 up to year 1
Population: 'Compliant-Use' set included PITT participants who completed at least one 28-day cycle and no other birth control methods were used. Cycles were excluded if a subject 1) skipped 2 or more consecutive combination pills, 2) had a pattern of substantial non-compliance with treatment, or 3) used a prohibited concomitant medication
Measure: Number (95% Confidence Interval); unit: pregnancies / 100 woman years exposure
Arm/Group | DR-103: Total | DR-103: <90 kg Subpopulation | DR-103: >=90kg Subpopulation
Number analyzed (Participants) | 2941 | 2531 | 531
pregnancies / 100 woman years exposure | 3.07 [2.3692 to 3.9105] | 2.68 [1.9696 to 3.5625] | 4.94 [2.9315 to 7.8034]

8. Primary Outcome: Summary of Participants With Treatment-emergent Adverse Events
Description: The on-treatment time frame spanned the time during which study drug was administered until 3 weeks beyond the last study drug date.
  Relationship to study drug was assessed by the investigator.
  Serious AEs (SAEs) are those that resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in an important medical event that may have jeopardized the patient or required medical or surgical intervention.
Time Frame: Day 1 up to 13 months
Population: Safety population of treated participants
Measure: Number; unit: participants
Arm/Group | DR-103
Number analyzed (Participants) | 3597
participants
  Treatment-emergent AEs (TEAEs) | 2605
  Treatment-related AEs | 1086
  Serious AEs | 58
  TEAEs leading to discontinuation | 463

9. Secondary Outcome: Compliant-Use Life-Table Estimates of Pregnancy Rates Based on 91-day Cycles and Broken Out by Subpopulations Defined by Participant Weight
Description: as for outcome 4
Time Frame: Day 1 up to year 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: pregnancies / cumulative exposure
Arm/Group | DR-103: Total | DR-103: <90 kg Subpopulation | DR-103: >=90kg Subpopulation
Number analyzed (Participants) | 2505 | 2067 | 438
pregnancies / cumulative exposure
  Cycle 1 | 0.0080 [0.0044 to 0.0144] | 0.0062 [0.0030 to 0.0130] | 0.0164 [0.0062 to 0.0431]
  Cycle 2 | 0.0134 [0.0083 to 0.0215] | 0.0116 [0.0066 to 0.0204] | 0.0215 [0.0090 to 0.0511]
  Cycle 3 | 0.0236 [0.0162 to 0.0344] | 0.0203 [0.0129 to 0.0317] | 0.0392 [0.0196 to 0.0776]
  Cycle 4 | 0.0291 [0.0206 to 0.0412] | 0.0256 [0.0170 to 0.0385] | 0.0457 [0.0238 to 0.0871]

ADVERSE EVENTS:
Time Frame: Day 1 - one year and three weeks
Arm/Group | DR-103
Serious Adverse Events (participants affected / at risk) | 58/3597
Other Adverse Events (participants affected / at risk) | 1567/3597
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DR-103 (N=3597)
Pneumonia (Infections and infestations) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Staphylococcal infection (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 5
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1
Pelvic inflammatory disease (Infections and infestations) | 1
Convulsion (Nervous system disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 2
Injury (Injury, poisoning and procedural complications) | 1
Atrial fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Convulsion (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Depression suicidal (Psychiatric disorders) | 1
Pharyngitis (Infections and infestations) | 1
Depression (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 5
Overdose (Injury, poisoning and procedural complications) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Hepatitis C (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Anxiety (Psychiatric disorders) | 1
Rectal abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 2
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1
Urinary tract infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Mental status changes (Psychiatric disorders) | 1
Pyelonephritis (Infections and infestations) | 2
Drug dependence (Psychiatric disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Salpingitis (Infections and infestations) | 1
Uterine inflammation (Reproductive system and breast disorders) | 1
Hip dysplasia (Congenital, familial and genetic disorders) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Ileitis (Gastrointestinal disorders) | 1
Helicobacter gastritis (Infections and infestations) | 1
Angina pectoris (Cardiac disorders) | 1
Multiple drug overdose (Injury, poisoning and procedural complications) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DR-103 (N=3597)
Nasopharyngitis (Infections and infestations) | 342
Upper respiratory tract infection (Infections and infestations) | 323
Sinusitis (Infections and infestations) | 246
Urinary tract infection (Infections and infestations) | 214
Metrorrhagia (Reproductive system and breast disorders) | 216
Dysmenorrhoea (Reproductive system and breast disorders) | 188
Nausea (Gastrointestinal disorders) | 241
Headache (Nervous system disorders) | 420
Acne (Skin and subcutaneous tissue disorders) | 193

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Details of the study and its results shall not be publicized or published in any form to cooperative publication without prior, written consent of sponsor. Such approval is necessary to prevent premature disclosure of trade secrets and other confidential information.